CLINICAL TRIAL: NCT04420754
Title: A Multicenter Phase I Study of AIC100 CAR T Cells in Relapsed and/or Refractory Advanced Thyroid Cancer or Anaplastic Thyroid Cancer
Brief Title: Study of AIC100 CAR T Cells in Relapsed/Refractory Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AffyImmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-12021154
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Anaplastic Thyroid Cancer; Relapsed/Refractory Poorly Differentiated Thyroid Cancer
Keywords: AIC100; CAR T Cell; Anaplastic Thyroid Cancer; Poorly Differentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort -1 (Experimental): AIC100 CAR T Cell Dose Level -1 (Flat Dose): 1 x 10e6 CAR T cells
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 1 (Experimental): AIC100 CAR T Cell Dose Level 1 (Flat Dose): 1 x 10e7 CAR T cells
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 2 (Experimental): AIC100 CAR T Cell Dose Level 2 (Flat Dose): 1 x 10e8 CAR T cells
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 3 (Experimental): AIC100 CAR T Cell Dose Level 3 (Flat Dose): 5 x 10e8 CAR T cells
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 2.5 (Experimental): AIC100 CAR T Cell Dose Level 2.5 (Flat Dose): 2.5 x 10e8 CAR T cells. The interim step-down dose of Cohort 2.5 may be evaluated, if needed, based on ongoing safety and efficacy data.
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 4 (Experimental): AIC100 CAR T Cell Dose Level 4 (Flat Dose): 7.5 x 10e8 CAR T cells. The proposed escalation dose of Cohort 4 may be evaluated, if needed, based on ongoing safety and efficacy data.
  Interventions: Biological: AIC100 CAR T Cells
- Cohort 5 (Experimental): AIC100 CAR T Cell Dose Level 5 (Flat Dose): 1 x 10e9 CAR T cells. The proposed escalation dose of Cohort 5 may be evaluated, if needed, based on ongoing safety and efficacy data.
  Interventions: Biological: AIC100 CAR T Cells

INTERVENTIONS:
Biological: AIC100 CAR T Cells — Autologous CAR T cells directed against ICAM-1
  Other Names: AIC100

SUMMARY:
The purpose of this study is to assess the safety and tolerability and determine the recommended Phase 2 dose of AIC100 Chimeric Antigen Receptor (CAR) T cells in patients with relapsed/refractory poorly differentiated thyroid cancer and anaplastic thyroid cancer, including newly diagnosed.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of AIC100 CAR T Cells and determine the recommended Phase 2 dose of AIC100 in patients with relapsed/refractory poorly differentiated thyroid cancer and in patients with anaplastic thyroid cancer that are BRAF wild-type, including newly diagnosed, or BRAF mutant anaplastic thyroid cancer after failure of BRAF mutant specific therapy.

Upon enrollment, patients will undergo apheresis for collection of autologous lymphocytes. The autologous T cells will be transfected and expanded in vitro to generate the AIC100 CAR T Cell product. After lymphodepleting chemotherapy, AIC100 CAR T Cells will be infused.

The study drug product, AIC100, consists of autologous CAR T cells targeting intercellular adhesion molecule-1 (ICAM-1) on thyroid cancer. In addition, AIC100 cells express the somatostatin receptor subtype 2 (SSTR2), which should enable imaging of AIC100 CAR T Cells.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate in the study and provide written informed consent
2. Be ≥ 18 years of age on the day of signing the Informed Consent Form
3. Patients must have thyroid cancer that meets one of the following diagnoses, and, prior to lymphodepleting chemotherapy (LDC), have an identified available fresh or archival biopsy sample:

   1. Anaplastic Thyroid Cancer BRAF wild-type at any stage, including newly diagnosed
   2. Anaplastic Thyroid Cancer BRAF mutant after failure of or inability to tolerate BRAF- specific therapy
   3. Poorly Differentiated Thyroid Cancer that has failed any of the following treatments: surgery radioactive iodine, chemotherapy, radiation therapy, and/or targeted therapies
4. Measurable disease by Computed Tomography (CT) or Positron Emission Tomography (PET) PET/CT per RECIST v1.1

   a. For ATC patients who do not have measurable disease at Screening, they are required to have measurable disease at Baseline Day -7 to proceed in the study.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
6. Life expectancy greater than 8 weeks
7. Overall adequate hepatic, renal, bone marrow, cardiac, and coagulation function, defined as the following:

   1. Estimated creatinine clearance ≥ 50 mL/minute
   2. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST): normal or Grade 1. Note: Lymphodepleting Chemotherapy (LDC) agents can cause fluctuations in hepatic enzymes.
   3. Serum total bilirubin: normal or Grade 1. Note: LDC agents can cause fluctuations in hepatic enzymes.
   4. Serum albumin: normal or Grade 1. (human albumin supplementation is not allowed within 2 weeks prior to Screening assessment)
   5. Hemodynamically stable and left ventricular ejection fraction ≥ 45%
   6. Hematological parameters

   i. Absolute neutrophil count > 1000/μL without myeloid growth factor support for ≥ 2 weeks

   ii. Absolute lymphocyte count ≥ 100/μL at screening and at apheresis

   iii. Platelet count ≥ 50 × 1000/μL without platelet transfusion for ≥ 2 weeks

   iv. Hemoglobin concentration > 7 g/dL without red blood cell transfusion for ≥ 2 weeks
8. Has met the minimum washout time for previous cancer treatments before undergoing apheresis or LDC, and in the Investigator's judgement, the patient is able to safely undergo the procedure
9. (incorporated into inclusion criteria #7)
10. Females of reproductive potential (defined as all females physiologically capable of becoming pregnant) must agree to use 1 highly effective method of contraception and 1 additional effective method from at least 30 days before enrollment/apheresis and for at least 1 year after the infusion of AIC100 CAR T Cells.
11. Females of reproductive potential must have a negative serum beta-human chorionic gonadotropin pregnancy test result at Screening

Exclusion Criteria:

1. Women who are pregnant or breastfeeding
2. Clinically significant, active, uncontrolled, systemic infection; the following are not exclusionary:

   1. Patients with Human immunodeficiency virus (HIV) must have been on effective antiretroviral therapy for ≥ 4 weeks prior to enrollment; must have an HIV viral load < 400 copies/µL; no acquired immunodeficiency syndrome related opportunistic infections in the previous 12 months; and a CD4+ cell count ≥ 350 cells/µL
   2. Patients with chronic hepatitis B virus (HBV) infection must be on antiviral therapy and have an HBV viral load below the limits of detection
   3. Patients with chronic hepatitis C virus (HCV) infection must have completed therapy and have an HCV viral load below the limits of detection
3. Prior treatment with investigational gene therapy or CAR T cell therapy
4. Presence of active and clinically relevant central nervous system disorder such as epilepsy, stroke, or symptomatic or uncontrolled brain metastases
5. Evidence of another malignancy within 2 years prior to Screening (except in-situ non melanoma skin cancers, localized controlled prostate cancer, adequately treated Stage 1 uterine cancer that has a low risk of recurrence, or any other malignancies with similar outcome)
6. (incorporated into exclusion criteria #2)
7. Active autoimmune disease (including but not limited to systemic lupus erythematosus, Sjögren's Syndrome, rheumatoid arthritis (RA), psoriasis, multiple sclerosis, inflammatory bowel disease) requiring immunosuppressive therapy within 4 weeks prior to eligibility confirmation
8. Patients with severe chronic diseases of the kidney, liver, heart, lung; or any other serious illness that, in the opinion of the Investigator, may affect the patient's treatment, follow up, or assessments, including but not limited to uncontrolled clinically significant neurological or psychiatric disorders or metabolic diseases
9. Patients who need long-term use of systemic corticosteroids > 10 mg/day prednisone or equivalent
10. Allergy to the chemotherapy drugs given during lymphodepletion or known hypersensitivity to any component of AIC100 CAR T Cells, including excipients
11. Receipt of a COVID-19 vaccine within 4 weeks before Screening
12. Concurrent participation in another interventional clinical study during participation in this study

    1. Prior treatment with any gene therapy or genetically modified cell therapy, including CAR T cells
    2. Prior treatment with ICAM-1 directed antibody, bispecific T cell engager, or antibody drug conjugate, unless there is confirmed ICAM-1 expression (by immunohistochemistry) after progression or relapse following most recent ICAM-1 directed treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2030-08-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of overall Grade >=3 Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 1 year post-infusion
  The number of Grade 3, 4 and 5 AEs and SAEs that occur throughout the study.
Incidence of anticipated AIC100 CAR T Cell related AEs, SAEs and adverse events of special interest (AESI) (infusion-related reactions, CRS, ICANS, HLH/MAS, TLS, new malignancies, AEs leading to death and DLT AEs) | Up to 15 years post-infusion
  The number of CAR T related adverse events that occur throughout the study, including AESIs, infusion-related reactions, cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS), tumor lysis syndrome (TLS) and new malignancies.
Determine recommended phase 2 dose | Up to 1 year post infusion
  The recommended phase 2 dose will be determined through the dose escalation process

SECONDARY OUTCOMES:
Assessment of presence and frequency of AIC100 CAR T cells in peripheral blood and tumor samples (when available) | Up to 15 years post-infusion
  Patients will be monitored for expansion and persistence of AIC100 CAR transgenes after infusion by vector copy number (VCN) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Gupta, MD PhD, Study Director — AffyImmune Therapeutics, Inc.
Locations (4):
- United States (4):
  - City of Hope National Medical Center, City of Hope Medical Center, Duarte, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No